CLINICAL TRIAL: NCT00689897
Title: Psychological Outcomes From a Study of Acupuncture Treatment on Experimentally Primary Dysmenorrhea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: The Fifth Hospital of Wuhan (Other)
Responsible Party: Psychological Outcomes From a Study of Acupuncture Treatment on Experimentally Primary Dysmenorrhea, Institute of Integrated Traditional Chinese and Western Medicine , Department of Neurology of Tongji Hospital，Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006CB504502-2
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-04

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Deqi; acupuncture; psychology
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): In acupuncture treatment, immediately after insertion of a needle, it is manually rotated backwards and forwards to induce the DeQi sensation, the needles are retained for 30 minutes.
  Interventions: Procedure: acupuncture, Deqi
- 2 (Active Comparator): In acupuncture treatment, immediately after insertion of a needle, it is NOT manually rotated backwards or forwards to induce the DeQi sensation, and retained for 30 minutes.
  Interventions: Procedure: acupuncture, Non-Deqi

INTERVENTIONS:
Procedure: acupuncture, Deqi — Immediately after insertion of a needle, it is manually rotated backwards and forwards to induce the DeQi sensation.
  Other Names: Deqi
  Arms: 1
Procedure: acupuncture, Non-Deqi — After insertion of a needle, no manipulation is applied, and the needle is retained for 30 minutes.
  Other Names: Non-Deqi
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the associations between deqi, the effects of acupuncture and personality in primary dysmenorrhea and to characterize the nature of the deqi phenomenon on terms of the prevalence of sensations as well as the uniqueness of the sensations underlying the deqi experiment.

DETAILED DESCRIPTION:
The mechanism, by which acupuncture works is not yet clear, therefore there is no unequivocal consensus about styles and sensations of acupuncture. whether psychological factor has influences on the effects of acupuncture? This study will adopt international practices such as visual analogue scale (VAS) to objective evaluation. The confident degree, feeling degree for acupuncture and pain intensity were evaluated by the patient with VAS, and the pain VAS scores before and after acupuncture were recorded as the indexes for assessment of the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age between 18 and 30 years old, who had regular menstrual cycles (28-33 days);
2. Meeting diagnostic criteria for primary dysmenorrhea, having moderate to severe symptoms when unmedicated, and eligible for care through the military health system.

Exclusion Criteria:

1. Secondary dysmenorrhea;
2. Women with systemic disease, or hormonal, psychiatric or gynecologic disorders, or substance abuse;
3. Pregnant or trying to conceive, using oral contraceptives, smoker, breast-feeding.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for pain intensity of primary dysmenorrhea | 90 days after onset

SECONDARY OUTCOMES:
average duration (hours) of pain | 90 days after onset

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Principal Investigator — Tongji Hospital
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Wuhan, Hubei, China